CLINICAL TRIAL: NCT06192758
Title: An Early Feasibility Study to Evaluate the Safety of the TheraSphere Prostate Cancer (PCa) Device in Patients With Clinically Localized Prostate Cancer
Brief Title: Dose Escalation Study Evaluating Safety of TheraSphere Prostate Cancer (PCa) Device
Acronym: VOYAGER
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to predetermined protocol stopping criteria
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S2493
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate; Cancer
Keywords: Radiation; TheraSphere; Y90; Yttrium-90; Glass; Microspheres
MeSH Terms: conditions — Neoplasms; Chromosome 2q32-Q33 Deletion Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will be treated in cohorts at three sequential target absorbed radiation dose levels, where the dose level for the next cohort will be determined by a prespecified decision tree for escalation/de-escalation, according to the accelerated Time-to-Event Bayesian Optimal Interval Design (TITE-BOIN) approach.
  * Cohort size = 3 subjects
  * ≤15 subjects (or 5 cohorts) will be treated at any single dose level. ≤ 36 subjects (or 12 cohorts) will be treated in total across all doses. If no dose limiting toxicities are observed at any dose level, a minimum of 21 subjects will be treated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TheraSphere PCa Dose Escalation (Experimental): Participants will be treated in cohorts of three across three sequential dose levels:
  * Dose Level 1 (or starting dose) = 175 Gy; however, a provisional lower dose level, Dose Level -1 = 150 Gy, may be utilized in case de-escalation is warranted at Dose Level 1.
  * Dose Level 2 = 200 Gy
  * Dose Level 3 = 225 Gy
  Interventions: Device: TheraSphere PCa

INTERVENTIONS:
Device: TheraSphere PCa — Single session treatment of TheraSphere PCa - Yttrium-90 Glass Microspheres for the treatment of prostate cancer. Dose vials will be available in activity ranging from 0.1 GBq (2.7 mCi) to 3 GBq (81 mCi).
  Other Names: TheraSphere PCa - Yttrium-90 Glass Microspheres

SUMMARY:
The VOYAGER Study is an interventional, non-randomized, single-arm, dose escalation trial with the goal of determining the safety of TheraSphere PCa device in patients with clinically localized prostate cancer across US-based centers.

DETAILED DESCRIPTION:
TheraSphere™ Y-90 Glass Microspheres are a targeted cancer therapy consisting of tiny glass beads containing radioactive Yttrium-90 (Y-90), which are injected directly into the blood vessel feeding the tumor through a microcatheter using advanced imaging guidance. The glass microspheres enter the tumor's blood supply, lodge within the blood vessels feeding the tumor, and release radiation to the tumor. The radiation works to destroy the tumor cells from within, thus limiting radiation exposure to surrounding normal tissues, a process referred to as selective internal radiation therapy (SIRT).

This study aims to investigate the maximum safe radiation dose of TheraSphere Prostate Cancer (PCa) device that can be delivered in patients with clinically localized prostate cancer. The study will also evaluate the full safety profile, technical feasibility, efficacy, and quality of life metrics of the TheraSphere PCa device.

Participants will be asked to complete the following:

* At least two image-guided visits, including a mapping assessment (without Technetium Tc albumin aggregated [Tc-MAA]) prior to treatment
* One treatment visit, including image-guided assessments
* Fifteen post-treatment follow-up visits for a total of approximately 20 visits over the 5-year study period

Note: the VOYAGER Study is a staged investigational device exemption (IDE) study; therefore, the full enrollment of 21 to 36 subjects is subject to FDA approval following safety review of the first 10 subjects enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has ability to comprehend and willingness to sign and date the IRB-approved study informed consent form (ICF), and to comply with the study testing, procedures, and follow-up schedule.
2. Histologic confirmation of adenocarcinoma of the prostate by MR-fusion biopsy. Referral biopsy for eligibility must be completed between 180 days and 6 weeks prior to mapping procedure.
3. Subject with favorable intermediate risk clinically localized prostate cancer defined per NCCN Guidelines version 3.2022 as follows:

   * Favorable intermediate-risk has all the following:
   * i. One Intermediate Risk Factor (IRF):

     1. cT2b-cT2c
     2. Grade Group 2 or 3
     3. PSA 10-20 ng/mL
   * ii. Grade Group 1 or 2
   * iii. <50% biopsy cores positive (e.g., <6 of 12 cores)
4. Staging MRI must confirm American Joint Committee on Cancer (AJCC, 8th edition) stage T1, T2a, T2b or T2c.
5. Whole prostate gland volume ≥ 60 cc (measured on MRI)
6. International Prostate Score Symptom (I-PSS) ≤ 18
7. Estimated life expectancy of >5 years according to NCCN guideline's tools (NCCN v03.2022) who has declined or is ineligible for Standard of Care treatments (observation, active surveillance, surgery, and radiation therapies [brachytherapy/external beam radiation therapy])
8. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
9. Angiographic inclusion criteria:

   * a. Type I to IV prostate artery origins on both hemiglands.1
   * b. No evidence of procedure limiting vascular abnormalities (aneurysms, stenosis, shunt, fistula, occlusion) or morphologic asymmetric single prostate artery on either side (hemigland)
   * c. Bilaterally accessible solitary prostatic arteries.
   * d. Complete perfusion of the prostate gland via a single dominant vessel for each hemigland
10. Have adequate organ and bone marrow function within 30 days prior to index procedure, as defined below:

    * a. International Normalized Ratio (INR) ≤ 1.2 (in absence of anticoagulation)
    * b. Platelets ≥ 75,000/L
    * c. GFR ≥ 40 mL/min/1.73m2
    * d. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
    * e. Hemoglobin (Hgb) ≥ 9.0 g/dL (Note: the use of transfusion or other intervention to achieve adequate bone marrow function is acceptable
    * f. ALT/AST ≤ 5 x upper limit of normal (ULN)
    * g. Bilirubin ≤ 2 mg/dL
11. Patients with known Human Immunodeficiency Virus (HIV) infection are eligible with well controlled HIV infection, no current or previous AIDS-related complications and CD4+ T-cell (CD4+) counts ≥ 350 cells/uL

Exclusion Criteria:

1. Direct evidence of regional or distant metastases after appropriate staging studies per NCCN guidelines (v03.2022)
2. Histological evidence of intraductal features
3. Previous treatments (pelvic radiotherapy, surgery, prostate artery embolization [PAE], transurethral resection of the prostate [TURP] or previous/ planned hormonal therapy
4. History of Crohn's Disease, ulcerative colitis, or ataxia telangiectasia, current gross haematuria, or current urinary catheter
5. Subjects with ongoing urinary tract infection, prostate abscess, prostatitis, or neurogenic bladder
6. Prior significant rectal surgery (haemorrhoidectomy is acceptable)
7. Prior invasive malignancy unless disease free for a minimum of 3 years. Exceptions to this requirement include adequately treated non-melanoma skin cancer or lentigo maligna or carcinoma in situ without evidence of disease
8. Hip prosthesis
9. Medical contraindication to undergo contrast-enhanced angiography, CT scan and magnetic resonance imaging (MRI), or arterial catheterization, or known history of hypersensitivity reactions to iodinated and gadolinium-based contrast product
10. Angiographic exclusion criteria:

    * a. Perfusion to tissues outside the Planning Target Volume (PTV) that cannot be corrected by placement of the catheter distal to collateral vessels or the application of standard angiographic techniques, such as coil embolization
    * b. Type V prostatic artery origin on either side

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated radiation dose of TheraSphere PCa | Through 90 days post-treatment
  • The Maximum Tolerated Dose (MTD) of Yttrium-90 Glass Microspheres (TheraSphere™ PCa) is based on rate of dose limiting toxicity (DLT) through 90 days, defined as any ≥ grade 3 adverse event (AE) according to CTCAE v.5

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Through 5 years post-treatment (acute ≤ 90 days and late > 90 days)
  The following AEs/SAEs will be assessed in accordance with National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0:
  * Rate of any ≥ grade 3 AEs
  * Rate of AEs of interest, i.e., any ≥ Grade 2 GI/GU and erectile dysfunction toxicities
  * Rate of any treatment-emergent AEs and treatment-emergent SAEs
  * Rate of any treatment-related AEs and treatment-related SAEs
  * AEs related to non-target TheraSphere PCa distribution
Rate of success of delivering intended dose | Immediately post-treatment
  • The ability to deliver the intended TheraSphere PCa absorbed dose (+/- 20%) to the treatment volume based on post-treatment PET derived absorbed dose.
Recurrence Free Survival | Through 5 years post-treatment
  • Biochemical Recurrence Free Survival (bRFS) based on PSA according to the Phoenix criteria (RTOG-ASTRO definition). Biochemical recurrence of prostate cancer after curative treatment is defined as a PSA rise of ≥ 2 ng/mL above the post-treatment nadir.
Progression free survival (PFS) | Through 5 years post-treatment
  • Progression free survival (PFS) and local progression free survival (LPFS), defined as time from inclusion until one of the following events, whichever comes first: biochemical progression (Phoenix criteria) or clinical progression.
Prostate cancer specific survival | Through 5 years post-treatment
  • Prostate cancer specific survival will be measured as the number of days between treatment with TheraSphere PCa and death by prostate cancer.
Overall survival (OS) | Through 5 years post-treatment
  • OS will be measured as the number of days between treatment with TheraSphere PCa and death by any cause.
Rate of subsequent prostate anticancer treatment | Through 5 years post-treatment
  • A summary table with number of subjects (%) who received subsequent definitive or systematic therapy and type of therapies received will be presented.
Rate of histopathological recurrence | Through 5 years post-treatment
  • Rate of recurrence based on histopathological assessment of prostate MR/US-fusion biopsy in patients with evidence of progression.
Quality of Life (QoL) measured by EPIC-26 | Through 5 years post-treatment
  • Change from baseline measured through Expanded Prostate Cancer Index Composite (EPIC-26).
Quality of Life (QoL) measured by MSHQ | Through 5 years post-treatment
  • Change from baseline measured through Male Sexual Health Questionnaire (MSHQ).
Quality of Life (QoL) measured by I-PSS | Through 5 years post-treatment
  • Change from baseline measured through International Prostate Symptom Score (I-PSS).
Maximum urinary flow (Qmax) | Through 5 years post-treatment
  • Change from baseline
Post-void residual (PVR) urine test | Through 5 years post-treatment
  • Change from baseline
Dose Distribution | Through one-week post-treatment
  • Dose Volume Histogram (DVH) and evaluation of D90 from post-treatment Y90 PET-MRI/CT.

OTHER OUTCOMES:
Prostatic imaging assessment | Through 5 years post-treatment
  • Qualitative analysis of multi-parametric MRI (mp-MRI) and PI-RADS score

CONTACTS AND LOCATIONS:
Overall Officials: Samdeep Mouli, M.D., M.S., Principal Investigator — Northwestern Medical Hospital; Mark Hurwitz, MD, Principal Investigator — Westchester Medical Center
Locations (5):
- United States (5):
  - Ronald Reagan UCLA Medical Center (UCLA Health, Los Angeles), Los Angeles, California
  - University of Miami (Sylvester Comprehensive Cancer Center), Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Mount Sinai Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mouli SK, Raiter S, Harris K, Mylarapu A, Burks M, Li W, Gordon AC, Khan A, Matsumoto M, Bailey KL, Pasciak AS, Manupipatpong S, Weiss CR, Casalino D, Miller FH, Gates VL, Hohlastos E, Lewandowski RJ, Kim DH, Dreher MR, Salem R. Yttrium-90 Radioembolization to the Prostate Gland: Proof of Concept in a Canine Model and Clinical Translation. J Vasc Interv Radiol. 2021 Aug;32(8):1103-1112.e12. doi: 10.1016/j.jvir.2021.01.282. Epub 2021 Apr 9. PMID 33839262
- [Background] Yuan Y, Lin R, Li D, Nie L, Warren KE. Time-to-Event Bayesian Optimal Interval Design to Accelerate Phase I Trials. Clin Cancer Res. 2018 Oct 15;24(20):4921-4930. doi: 10.1158/1078-0432.CCR-18-0246. Epub 2018 May 16. PMID 29769209
- [Derived] Meiselman S, Thomas MA, Giardina JD, Zheleznyak A, Thorek DLJ, Malone CD. Advances in Radioembolization for Liver Cancer. J Vasc Interv Radiol. 2025 Dec;36(12):1876-1881. doi: 10.1016/j.jvir.2025.07.018. PMID 41276366